CLINICAL TRIAL: NCT04566731
Title: Using Transcranial Direct Current Stimulation to Reveal Mechanisms of Language Loss and to Treat Progressive Aphasia Associated With FTD and Related Dementias
Brief Title: Treating Primary Progressive Aphasia (PPA) Using tDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 843286
Record Dates: First submitted 2020-08-31; First posted 2020-09-28 (Actual); Results first posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Primary Progressive Aphasia
Keywords: non-invasive brain stimulation; transcranial direct current stimulation (tDCS); speech therapy
MeSH Terms: conditions — Aphasia, Primary Progressive; Communication Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Crossover assignment
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- tDCS + CILT (Active Comparator): Participants will undergo 10 daily sessions (Monday-Friday, x2 weeks) of tDCS for 20 minutes using a montage in which an anode (1.5 mA) is placed over F7 (left frontotemporal lobe) and the cathode will be place on O1 (left occipital) using the 10-20 EEG mapping system. Subjects will participate in a modified constraint-induced language therapy.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS); Behavioral: Modified Contraint-Induced Language Therapy (mCILT)
- Sham tDCS + CILT (Sham Comparator): Participants will undergo 10 daily sessions (Monday-Friday, x2 weeks) of sham tDCS for 20 minutes using a montage in which an anode is placed of F7 and cathose is placed over O1. Subjects will participate in a modified constraint-induced language therapy,
  Interventions: Device: Sham tDCS; Behavioral: Modified Contraint-Induced Language Therapy (mCILT)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — tDCS is a type of non-invasive brain stimulation in which small electrical currents are applied to the scalp via 2 electrodes. The current, 1.5 mA, is approximately of the same intensity as the current provided by a 9-volt battery. To deliver the current, electrodes that are placed in saline soaked sponges. They will be attached to the left side of your head; they will be held in place with an elastic cap. For both real and sham stimulation the electrodes will be placed on the scalp.
  Arms: tDCS + CILT
Device: Sham tDCS — tDCS is a type of non-invasive brain stimulation in which small electrical currents are applied to the scalp via 2 electrodes. During sham stimulation, the current, 1.5 mA, will be delivered for a short amount of time and then turn-off. To deliver the current, electrodes that are placed in saline soaked sponges. They will be attached to the left side of your head; they will be held in place with an elastic cap. For both real and sham stimulation the electrodes will be placed on the scalp. Most people cannot tell the difference between real and sham stimulation.
  Arms: Sham tDCS + CILT
Behavioral: Modified Contraint-Induced Language Therapy (mCILT) — Modified constraint-induced language therapy (mCILT) is a behavioral language therapy that invokes use-dependent learning in communicative interactions by requiring spoken output and restricting use of alternative forms of communication, such as gestures, as a substitute for spoken output. Other key elements of CILT include massed practice of goal-directed speech and shaping of desired responses by increasing response demands as participants improve. MCILT differs from traditional constraint-induced language therapy (CILT) in three ways: 1) it will be done as an individual therapy with the examiner in the role of a communication partner; 2) treatment will be delivered in short sessions (1 hour rather than a more typical 3-4 hour session); 3) targeting nouns + semantically related verbs to generate noun + verb phrases in treatment, a modification that may be better suited to addressing syntactic structure.

SUMMARY:
This is a double-blind, sham-controlled, crossover study in which subjects with the non-fluent/agrammatic and semantic variants of primary progressive aphasia (naPPA and svPPA, respectively) will undergo language testing and structural and functional brain imaging before and after receiving 10 semi-consecutive daily sessions of real or sham transcranial direct current stimulation (tDCS) paired with modified constraint-induced language therapy (mCILT). Language testing and brain imaging will be repeated immediately after completion of and up-to 24 weeks following completion of treatment. The investigators will examine changes in language performance induced by tDCS + mCILT compared to sham tDCS + mCILT. The investigators will also use network science to analyze brain imaging (fMRI) data to identify network properties associated with baseline PPA severity and tDCS-induced changes in performance. This study will combine knowledge gained from our behavioral, imaging, and network data in order to determine the relative degrees to which these properties predict whether persons with PPA will respond to intervention.

DETAILED DESCRIPTION:
The central framework for the project is a double-blind, sham-controlled, crossover study in which subjects with the non-fluent/agrammatic and semantic variants of primary progressive aphasia (naPPA and svPPA, respectively) will undergo language testing and structural and functional brain imaging before and after receiving 10 semi-consecutive daily sessions of real or sham transcranial direct current stimulation (tDCS) paired with modified constraint-induced language therapy (mCILT). Language testing and brain imaging will be repeated immediately after completion of and up-to 24 weeks following completion of treatment.

Subjects with naPPA and svPPA will be randomized to one of two study arms: tDCS+mCILT or sham stimulation+mCILT paired with pre- and post-stimulation imaging and behavioral measures. Equal numbers of subjects with naPPA and svPPA will be randomized to the tDCS + mCILT and sham + mCILT study arms. The study is double-blinded, in that neither the subject nor the study personnel administering tDCS or sham stimulation will know which arm of the study the subject has been randomized into. Study coordinators will administer tDCS by entering a pre-determined code that has been programmed into the device by another member of the study team. Data will be digitally audio-recorded and analyzed off-line, such that study team members performing data coding and analysis will likewise be blinded to the treatment condition of each subject.

Subject participation in this protocol will occur during 36 planned visits that will span approximately 12 months. The events of the study visits are described below:

VISIT 1:

Informed consent and screening

VISIT 2:

Baseline MRI

VISIT 3 & 4:

Baseline language assessment

VISITS 5-14:

tDCS+mCILT OR sham stimulation+mCILT, depending on the study arm to which they had been randomized.

VISIT 15 & 16:

Follow-up language assessment Follow-up MRI

VISIT 17:

6-Week follow-up language assessment

VISIT 18 & 19:

12-week follow-up language assessment 12-week follow-up MRI

**CROSSOVER**

VISIT 20:

Crossover baseline language assessment

VISITS 21-30:

tDCS+mCILT or sham stimulation+mCILT

VISIT 31 & 32:

Follow-up language assessment Follow-up MRI

VISIT 33:

6 Week follow-up language assessment

VISIT 34 & 35:

12-week follow-up language assessment 12-week follow-up MRI

VISIT 36:

24 week follow-up language assessment

ELIGIBILITY:
Inclusion Criteria:

* Presence of aphasia attributable to the semantic variant (svPPA) or non- fluent/agrammatic variant (naPPA) of Primary Progressive Aphasia.
* Must be a native English speaker

Exclusion Criteria:

* History of seizures or unexplained loss of consciousness
* Subjects with metallic objects in the face or head other than dental apparatus such as braces, ﬁllings, and implants.
* Subjects with Pacemakers or ICDs.
* Subjects with previous craniotomy or any breach in the skull
* Subjects with a history of other neurological disorder (stroke, TBI, Parkinson)
* Subjects with a history of small vessel disease

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Hamilton, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from July 2020-July 2024 from the Hospital of the University of Pennsylvania and surrounding Philadelphia area medical centers.
Pre-assignment Details: A total of 3 participants did not qualify at the time of enrollment due to low MMSE scores (2) and diagnosis change that no longer met our PPA criteria (1).
  A total of 2 participants dropped out of the study before they were randomized due to travel concerns.
Groups:
- tDCS + CILT First, Then Sham tDCS + CILT: Participants will undergo 10 daily sessions (Monday-Friday, x2 weeks) of tDCS for 20 minutes using a montage in which an anode (1.5 mA) is placed over F7 (left frontotemporal lobe) and the cathode will be place on O1 (left occipital) using the 10-20 EEG mapping system. Subjects will simultaneously participate in a modified constraint-induced language therapy.
  Follow-up language assessments will be completed immediately, 6 weeks and 12 weeks after tDCS + CILT treatment.
  After a 12 week washout period, participants will then crossover to the Sham tDCS condition. Follow-up language assessments will be completed immediately, 6 weeks,12 weeks and 24 weeks after Sham tDCS + CILT treatment.
- Sham tDCS + CILT First, Then tDCS + CILT: Participants will undergo 10 daily sessions (Monday-Friday, x2 weeks) of sham tDCS for 20 minutes using a montage in which an anode is placed of F7 and cathode is placed over O1. During sham stimulation, the current, 1.5 mA, will be delivered for a short amount of time (about 30 seconds) and then turn-off. Most people cannot tell the difference between real and sham stimulation. Subjects will simultaneously participate in a modified constraint-induced language therapy.
  Follow-up language assessments will be completed immediately, 6 weeks and 12 weeks after Sham tDCS + CILT treatment.
  After a 12 week washout period, participants will then crossover to the tDCS condition. Follow-up language assessments will be completed immediately, 6 weeks,12 weeks and 24 weeks after tDCS + CILT treatment.
Period: Overall Study
Arm/Group | tDCS + CILT First, Then Sham tDCS + CILT | Sham tDCS + CILT First, Then tDCS + CILT
Started | 10 | 8
Completed | 9 | 4
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- tDCS + CILT First, Then Sham + CILT: Participants will undergo 10 daily sessions (Monday-Friday, x2 weeks) of tDCS for 20 minutes using a montage in which an anode (1.5 mA) is placed over F7 (left frontotemporal lobe) and the cathode will be place on O1 (left occipital) using the 10-20 EEG mapping system. Subjects will simultaneously participate in a modified constraint-induced language therapy.
  Participants will then crossover to the Sham tDCS condition.
- Sham tDCS + CILT First, Then tDCS + CILT: Participants will undergo 10 daily sessions (Monday-Friday, x2 weeks) of sham tDCS for 20 minutes using a montage in which an anode is placed of F7 and cathode is placed over O1. During sham stimulation, the current, 1.5 mA, will be delivered for a short amount of time (about 30 seconds) and then turn-off. Most people cannot tell the difference between real and sham stimulation. Subjects will simultaneously participate in a modified constraint-induced language therapy.
  Participants will then crossover into the tDCS condition.
- Total: Total of all reporting groups
Arm/Group | tDCS + CILT First, Then Sham + CILT | Sham tDCS + CILT First, Then tDCS + CILT | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (5.89) | 68 (6.65) | 67.7 (6.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 8 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 8 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Western Aphasia Battery (WAB-AQ) Score [Mean (Standard Deviation); unit: scores on a scale] | 74.9 (12.84) | 78.0 (13.48) | 76.3 (13.2)

OUTCOME MEASURES:

1. Primary Outcome: Western Aphasia Battery Aphasia Quotient (WAB-AQ)
Description: The primary outcome measure will be the change in score on the Western Aphasia Battery Aphasia Quotient (WAB-AQ), a score assessing overall aphasia recovery. Scores can range from 0-100, with higher scores representing better outcomes. 0-25 is very severe, 26-50 is severe, 51-75 is moderate, and 76-above is mild. A score of 93 or higher is considered recovered.
Time Frame: Baseline to 12 weeks; baseline to 24 weeks when available
Population: 24 week follow-up data are not available for individuals randomized to the tDCS + CILT first, then Sham tDCS + CILT group because there is no 24 week follow-up for the first arm. 24 week follow-up data are not available for individuals randomized to the Sham tDCS + CILT first, then tDCS + CILT group because there is no 24 week follow-up for the first arm.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- tDCS + CILT First, Then Sham tDCS + CILT: Participants will undergo 10 daily sessions (Monday-Friday, x2 weeks) of tDCS for 20 minutes using a montage in which an anode (1.5 mA) is placed over F7 (left frontotemporal lobe) and the cathode will be place on O1 (left occipital) using the 10-20 EEG mapping system. Subjects will simultaneously participate in a modified constraint-induced language therapy.
  Participants will then crossover to the Sham tDCS condition.
Arm/Group | tDCS + CILT First, Then Sham tDCS + CILT | Sham tDCS + CILT First, Then tDCS + CILT
Number analyzed (Participants) | 9 | 5
scores on a scale
  tDCS: Baseline | 74.4 (14.2) | 76.5 (12.5)
  tDCS: 12 Week Follow-up | 72.5 (15.9) | 76.0 (15.9)
  Sham: Baseline | 72.5 (15.9) | 80.7 (9.0)
  Sham: 12 Week Follow-up | 72.2 (17.6) | 76.5 (12.5)
  Active: 24 Week Follow-up: number analyzed (Participants) | 0 | 5
  Active: 24 Week Follow-up |  | 75.0 (15.9)
  Sham: 24 Week Follow-up: number analyzed (Participants) | 9 | 0
  Sham: 24 Week Follow-up | 67.5 (21.1) |
Statistical Analysis 1: Comparison: tDCS + CILT First, Then Sham tDCS + CILT vs Sham tDCS + CILT First, Then tDCS + CILT; Test type: Superiority; p < .05, ANOVA

ADVERSE EVENTS:
Time Frame: From baseline, adverse event data were collected over a period of time consisting of 36 weeks (12 weeks for arm 1 and 24 weeks for arm 2).
Description: Adverse event (AEs) information was collected daily during treatment sessions, as well as each follow-up visit.
  This is a crossover study, meaning all participants received the real intervention at some point during their participation.
Groups:
- tDCS + CILT: Participants will undergo 10 daily sessions (Monday-Friday, x2 weeks) of tDCS for 20 minutes using a montage in which an anode (1.5 mA) is placed over F7 (left frontotemporal lobe) and the cathode will be place on O1 (left occipital) using the 10-20 EEG mapping system. Subjects will simultaneously participate in a modified constraint-induced language therapy.
  Follow-up language assessments will be completed immediately, 6 weeks and 12 weeks after treatment.
- Sham tDCS + CILT: Participants will undergo 10 daily sessions (Monday-Friday, x2 weeks) of sham tDCS for 20 minutes using a montage in which an anode is placed of F7 and cathode is placed over O1. During sham stimulation, the current, 1.5 mA, will be delivered for a short amount of time (about 30 seconds) and then turn-off. Most people cannot tell the difference between real and sham stimulation. Subjects will simultaneously participate in a modified constraint-induced language therapy.
  Follow-up language assessments will be completed immediately, 6 weeks and 12 weeks after treatment.
Arm/Group | tDCS + CILT | Sham tDCS + CILT
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/18 | 1/18
Other Adverse Events (participants affected / at risk) | 4/18 | 3/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tDCS + CILT (N=18) | Sham tDCS + CILT (N=18)
Hip replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tDCS + CILT (N=18) | Sham tDCS + CILT (N=18)
skin irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Fall (General disorders) | 1 (1) | 1 (1)
Headache (General disorders) | 1 (2) | 0 (0)
ear biopsy (Surgical and medical procedures) | 0 (0) | 1 (1)
Macular Degeneration (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/31/NCT04566731/Prot_SAP_000.pdf